CLINICAL TRIAL: NCT02825862
Title: Circumventing the 'Ick' Factor: a Multi-site Randomised Trial of the Effects of Omitting Affective Attitudes to Increase Intention to Become an Organ Donor
Brief Title: Investigating Affective Attitude Question-behaviour Effects on Intention to Become an Organ Donor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: University of Stirling (Other); Manipal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: REC1048b
Record Dates: First submitted 2016-06-14; First posted 2016-07-07 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2018-04

CONDITIONS: Organ Donation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Replication group (No Intervention): Replication group - this group will complete the entire questionnaire, in order to replicate the findings of O'Carroll et al (2011)
- Omit affective attitudes (Active Comparator): Omitting affective attitudes The intervention is the omission of all questions on affective attitudes. This group will complete a similar questionnaire to the replication group, with the same number of questionnaire items, but affective attitudes will be omitted. Dummy questions (e.g. about politics) will be substituted for these deleted questions.
  Interventions: Behavioral: Question-behaviour effect (for affective attitudes)
- Omit negatively-worded items (Active Comparator): Omitting negatively-worded affective attitudes. This intervention is the omission of a subset of negatively-worded affective attitudinal items. This group will complete a similar questionnaire to the replication group, with the same number of items, but all negatively-worded affective attitudes will be omitted. Dummy questions (e.g. about politics) will be substituted for these deleted questions.
  Interventions: Behavioral: Question-behaviour effect (negatively-worded attitudes)

INTERVENTIONS:
Behavioral: Question-behaviour effect (for affective attitudes) — Investigators propose to investigate the Question-behaviour effect (omit affective attitudes). Investigators will conduct an experimental manipulation by omitting certain items from a questionnaire assessing attitudes to organ donation. Specifically, investigators will omit questions on affective attitudes. This group will complete a similar questionnaire to the comparison group, with the same number of items, but items on affective attitudes will substituted for non-affective items (e.g. on political parties).
  Other Names: Priming
  Arms: Omit affective attitudes
Behavioral: Question-behaviour effect (negatively-worded attitudes) — Behavioral: Question-behaviour effect (for negatively-worded attitudes) Investigators propose to investigate the Question-behaviour effect (omit negatively-worded affective attitudes). Investigators will conduct an experimental manipulation by omitting certain items from a questionnaire assessing attitudes to organ donation. Specifically, investigators will omit questions on negatively-worded affective attitudes. This group will complete a similar questionnaire to the comparison group, with the same number of items, but items on negatively-worded affective attitudes will substituted for non-affective items (e.g. on political parties).
  Other Names: Priming
  Arms: Omit negatively-worded items

SUMMARY:
The investigators aim to experimentally manipulate presence of questions on positive or negative affective attitudes to see if including these moderate as intention to become an organ donor. The methodology will be replicated across three international sites (RCSI Dublin, RCSI Bahrain, RCSI Perdana University).

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate

Exclusion Criteria:

* Refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 999 (Actual)
Dates: Start 2016-02; Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Intention to become an organ donor | within 3 months
  Mean score of two 7-point items: "I will definitely sign up for organ donation and discuss this with my family in the next few months" and "How strong is your intention to sign up for organ donation and discuss this with my family in the next few months?"

SECONDARY OUTCOMES:
Taking a donor card after the interview | Immediately at the end of the interview (i.e. that day, an average of 10-15 minutes after consenting to participate))
  "Did survey participant accept a donor card?" Yes/No

CONTACTS AND LOCATIONS:
Overall Officials: Frank Doyle, PhD, Principal Investigator — Royal College of Surgeons in Ireland
Locations (4):
- Manipal University, Manipal, Karnataka, India
- RCSI, Dublin, Ireland
- RCSI Perdana University, Perdana, Serdang, Malaysia
- University of Stirling, Stirling, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided